CLINICAL TRIAL: NCT01271803
Title: A Phase IB, Open-Label, Dose-Escalation Study Evaluating the Safety, Tolerability and Pharmacokinetics of Vemurafenib in Combination With GDC-0973 (Cobimetinib) When Administered in BRAFV600E Mutation-Positive Patients Previously Treated (But Without Prior Exposure to BRAF or MEK Inhibitor Therapy) or Previously Untreated for Locally Advanced/Unresectable or Metastatic Melanoma or Those Who Have Progressed After Treatment With Vemurafenib
Brief Title: A Study of Vemurafenib and GDC-0973 (Cobimetinib) in Participants With BRAFV600E Mutation-Positive Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO25395
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Results first posted 2016-06-17 (Estimated); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — cobimetinib; Vemurafenib

ARMS (12):
- DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib (Experimental): Participants will receive oral 60 milligrams (mg) cobimetinib once daily (QD) on Days 1-14, followed by 14 days off on Days 15-28 (14/14 dosing schedule) and oral 720 mg vemurafenib twice daily (BID) on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: Cobimetinib; Drug: vemurafenib
- DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib (Experimental): Participants will receive oral 60 mg cobimetinib QD on Days 1-21, followed by 7 days off on Days 22-28 (21/7 dosing schedule) and oral 720 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: Cobimetinib; Drug: vemurafenib
- DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib (Experimental): Participants will receive oral 60 mg cobimetinib QD on 21/7 dosing schedule and oral 960 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: Cobimetinib; Drug: vemurafenib
- DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib (Experimental): Participants will receive oral 60 mg cobimetinib QD on Days 1-28 (28/0 dosing schedule) and oral 720 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: Cobimetinib; Drug: vemurafenib
- DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib (Experimental): Participants will receive oral 60 mg cobimetinib QD on 28/0 dosing schedule and oral 960 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: Cobimetinib; Drug: vemurafenib
- DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib (Experimental): Participants will receive oral 80 mg cobimetinib QD on 14/14 dosing schedule and oral 720 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: Cobimetinib; Drug: vemurafenib
- DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib (Experimental): Participants will receive oral 100 mg cobimetinib QD on 14/14 dosing schedule and oral 720 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: Cobimetinib; Drug: vemurafenib
- DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib (Experimental): Participants will receive oral 60 mg cobimetinib QD on 14/14 dosing schedule and oral 960 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: Cobimetinib; Drug: vemurafenib
- DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib (Experimental): Participants will receive oral 80 mg cobimetinib QD on 14/14 dosing schedule and oral 960 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: Cobimetinib; Drug: vemurafenib
- Cobimetinib Monotherapy (100 mg or 60 mg) (Experimental): Participants will receive oral 60 mg cobimetinib QD on 21/7 dosing schedule, or oral 100 mg cobimetinib QD on 14/14 dosing schedule of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: Cobimetinib
- CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib (Experimental): Participants will receive oral 60 mg cobimetinib QD on 21/7 dosing schedule and oral 720 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: Cobimetinib; Drug: vemurafenib
- CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib (Experimental): Participants will receive oral 60 mg cobimetinib QD on 21/7 dosing schedule and oral 960 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Interventions: Drug: Cobimetinib; Drug: vemurafenib

INTERVENTIONS:
Drug: Cobimetinib — Participants will receive cobimetinib 60 to 100 mg at any of the 3 dosing schedules with or without vemurafenib in cycles of 28 days each until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Other Names: GDC-0973
Drug: vemurafenib — Participants will receive vemurafenib 720 or 960 mg along with cobimetinib in cycles of 28 days each until disease progression, unacceptable toxicity, or any other discontinuation criteria are met.
  Arms: CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib; CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib; DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib; DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib; DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib; DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib; DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib; DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib; DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib; DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib; DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib

SUMMARY:
This open-label, dose-escalation study of vemurafenib in combination with cobimetinib will evaluate the safety, tolerability and pharmacokinetics in participants with BRAFV600 mutation-positive metastatic melanoma. Participants with previously untreated, BRAFV600E mutation-positive, locally advanced/unresectable or metastatic melanoma or those who have progressed on vemurafenib monotherapy immediately prior to enrolling in this trial are eligible. Participants will be assigned to different cohorts with escalating oral doses of vemurafenib and cobimetinib. This study consists of 2 stages, Stage 1 (Dose Escalation Stage [DES] and Cohort Expansion Stage [CES]) and the anticipated time on study treatment is until disease progression, unacceptable toxicity or any other discontinuation criterion is met.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically confirmed melanoma (unresectable Stage IIIc and Stage IV metastatic melanoma, as defined by American Joint Committee on Cancer [AJCC])
* Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) Version (V) 1.1
* Eastern Cooperative Oncology Group (ECOG) Performance Status of less than or equal to (</=) 1
* Participants must

  1. be previously untreated for locally advanced/unresectable or metastatic melanoma or
  2. previously treated but without prior exposure to any BRAF or MEK inhibitor therapy or
  3. progressed on vemurafenib while participating in a Phase I (including clinical pharmacology studies), II, or III clinical study or expanded access programs (EAP) immediately prior to enrollment in this study or
  4. progressed on vemurafenib administered in a postmarketing setting immediately prior to enrollment in this study.
* Life expectancy >/=12 weeks

Exclusion Criteria:

* History of prior significant toxicity from another RAF or MEK pathway inhibitor requiring discontinuation of treatment
* Palliative radiotherapy within 2 weeks prior to first dose of study drug treatment
* Experimental therapy within 4 weeks prior to first dose of study drug treatment except vemurafenib
* Major surgery within 4 weeks of first dose of study drug treatment or planning a major surgery during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-02-17 (Actual); Primary Completion 2013-10-01 (Actual); Study Completion 2017-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- United States (9):
  - UCLA Department of Medicine, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - The Angeles Clinic and Research Institute, Santa Monica Office, Santa Monica, California
  - University of Colorado; Anschutz Cancer Pavilion, Aurora, Colorado
  - University of Chicago, Chicago, Illinois
  - Indiana University - Department of Medicine, Division of Gastroenterology/Hepatology, Indianapolis, Indiana
  - Karmanos Cancer Inst. ; Hudson Webber; Cancer Research Building, Detroit, Michigan
  - New York University Medical Center, New York, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Peter Maccallum Cancer Institute; Medical Oncology, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Ascierto PA, Ribas A, Larkin J, McArthur GA, Lewis KD, Hauschild A, Flaherty KT, McKenna E, Zhu Q, Mun Y, Dreno B. Impact of initial treatment and prognostic factors on postprogression survival in BRAF-mutated metastatic melanoma treated with dacarbazine or vemurafenib +/- cobimetinib: a pooled analysis of four clinical trials. J Transl Med. 2020 Aug 3;18(1):294. doi: 10.1186/s12967-020-02458-x. PMID 32746839
- [Derived] Ribas A, Gonzalez R, Pavlick A, Hamid O, Gajewski TF, Daud A, Flaherty L, Logan T, Chmielowski B, Lewis K, Kee D, Boasberg P, Yin M, Chan I, Musib L, Choong N, Puzanov I, McArthur GA. Combination of vemurafenib and cobimetinib in patients with advanced BRAF(V600)-mutated melanoma: a phase 1b study. Lancet Oncol. 2014 Aug;15(9):954-65. doi: 10.1016/S1470-2045(14)70301-8. Epub 2014 Jul 15. PMID 25037139
- [Derived] Baudy AR, Dogan T, Flores-Mercado JE, Hoeflich KP, Su F, van Bruggen N, Williams SP. FDG-PET is a good biomarker of both early response and acquired resistance in BRAFV600 mutant melanomas treated with vemurafenib and the MEK inhibitor GDC-0973. EJNMMI Res. 2012 May 31;2(1):22. doi: 10.1186/2191-219X-2-22. PMID 22651703

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study included two stages. Stage 1: dose escalation stage (DES), consisted of 9 "Cobimetinib + Vemurafenib" combination arms and 1 Cobimetinib monotherapy. Stage 2: cohort expansion stage (CES), consisted of 2 "Cobimetinib + Vemurafenib" combination arms, treated with recommended phase 2 dose.
Pre-assignment Details: Participants data were pooled across dose/regimen cohorts from two stages and analyzed separately per final analysis for vemurafenib-PD and BRAFi-naive participants who received cobimetinib and vemurafenib. Data is presented based on the final CSR. As of 2017 per-cohort data were not collected
Groups:
- Vemurafenib PD Participants: All participants who progressed on vemurafenib monotherapy immediately prior to enrollment into this study were treated with vemurafenib in combination with cobimetinib at a particular dose combination and dosing schedule depending on the cohort in which they were enrolled until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- BRAFi-naïve Participants: All participants who were previously untreated or previously treated but naïve to BRAF or MEK inhibitor therapy were considered as BRAFi-naïve participants. These participants were treated with vemurafenib in combination with cobimetinib at a particular dose combination and dosing schedule depending on the cohort in which they were enrolled until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
- Cobimetinib Monotherapy (100 mg or 60 mg): Participants received oral 60 mg cobimetinib QD on 21/7 dosing schedule, or oral 100 mg cobimetinib QD on 14/14 dosing schedule of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
Period: Overall Study
Arm/Group | Vemurafenib PD Participants | BRAFi-naïve Participants | Cobimetinib Monotherapy (100 mg or 60 mg)
Started | 66 | 63 | 2
Completed | 11 | 24 | 0
Not Completed | 55 | 39 | 2
Not completed — Progressive disease | 0 | 0 | 2
Not completed — Death | 53 | 34 | 0
Not completed — Withdrawal by Subject | 1 | 5 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Demographic data was not reported across dose/regimen cohort per final analysis, as it was pooled across separately for vemurafenib-PD and BRAFi-naive participants who received cobimetinib and vemurafenib. Data is presented based on the final CSR. As of 2017 per-cohort data were not collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Vemurafenib PD Participants | BRAFi-naïve Participants | Cobimetinib Monotherapy (100 mg or 60 mg) | Total
Number analyzed (Participants) | 66 | 63 | 2 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (14.8) | 54.0 (13.0) | 62.5 (9.2) | 53.6 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 1 | 53
  Male | 42 | 35 | 1 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) During DES in Combination Cohorts
Description: DLT is defined as 1 of the following toxicities considered by the investigator to be related to study treatment: a) Grade 3 nausea, vomiting or diarrhea that resolved to Grade less than or equal to (≤) 1 within 7 days, b) Grade 3 rash or photosensitivity that resolved to Grade ≤2 within 7 days, c) Grade 3 cutaneous squamous cell carcinoma (cuSCC) that was subsequently resected, d) Grade greater than or equal to (≥) 3 fatigue or hyperuricemia that resolved to Grade ≤2 within 7 days, e) Grade 3 fever, f) Grade 3 or 4 elevation of serum creatine phosphokinase (CPK) levels, which is asymptomatic, deemed by the investigator to be clinically insignificant and that returned to Grade ≤2 during the 14-day cobimetinib treatment holiday, g) Grade ≥3 febrile neutropenia, h) Grade ≥4 neutropenia (absolute neutrophil count [ANC] less than <500/microliter [μL]), i) Grade ≥4 thrombocytopenia, j) Grade ≥4 anemia, k) Grade ≥3 elevation of total bilirubin, hepatic transaminase or alkaline phosphatase.
Time Frame: 28 Days
Population: Safety-evaluable population (SEP) included all participants who received at least one dose of study drug. SEP participants who received combination study treatment (cobimetinib + Vemurafenib) were included in the analysis of this outcome. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: participants
Groups:
- DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib: Participants received oral 60 mg cobimetinib QD on 14/14 dosing schedule and oral 720 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib: Participants received oral 60 mg cobimetinib QD on 21/7 dosing schedule and oral 720 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib: Participants received oral 60 mg cobimetinib QD on 21/7 dosing schedule and oral 960 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib: Participants received oral 60 mg cobimetinib QD on 28/0 dosing schedule and oral 720 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib: Participants received oral 60 mg cobimetinib QD on 28/0 dosing schedule and oral 960 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib: Participants received oral 80 mg cobimetinib QD on 14/14 dosing schedule and oral 720 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib: Participants received oral 100 mg cobimetinib QD on 14/14 dosing schedule and oral 720 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib: Participants received oral 60 mg cobimetinib QD on 14/14 dosing schedule and oral 960 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib: Participants received oral 80 mg cobimetinib QD on 14/14 dosing schedule and oral 960 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
Arm/Group | DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 5 | 8 | 27 | 3 | 4 | 4 | 4 | 3 | 5
participants | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1

2. Primary Outcome: Maximum Tolerated Doses (MTD) of Vemurafenib and Cobimetinib When Administered in Combination in DES
Description: The highest dose level(s) at which fewer than one-third of participants experienced a DLT was declared the MTD. DLT is defined as 1 of the following toxicities considered by the investigator to be related to study treatment: a) Grade 3 nausea, vomiting or diarrhea that resolved to Grade ≤1 within 7 days, b) Grade 3 rash/photosensitivity that resolved to Grade ≤2 within 7 days, c) Grade 3 cuSCC that was subsequently resected, d) Grade ≥3 fatigue/hyperuricemia that resolved to Grade ≤2 within 7 days, e) Grade 3 fever, f) Grade 3 or 4 elevation of serum CPK levels, which is asymptomatic, deemed to be clinically insignificant and returns to Grade ≤2 during the 14-day cobimetinib treatment holiday, g) Grade ≥3 febrile neutropenia, h) Grade ≥4 neutropenia (ANC <500/ μL), i) Grade ≥4 thrombocytopenia, j) Grade ≥4 anemia, k) Grade ≥3 elevation of total bilirubin, hepatic transaminase or alkaline phosphatase.
Time Frame: 28 Days
Population: Safety-evaluable population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Number; unit: mg
Groups:
- Dose Escalation Stage (Stage 1): All participants who received vemurafenib and cobimetinib in any dose combination during DES, until disease progression, unacceptable toxicity, or any other discontinuation criterion was met.
Arm/Group | Dose Escalation Stage (Stage 1)
Number analyzed (Participants) | 63
mg
  Cobimetinib dose (21/7 dosing schedule) | 60
  Vemurafenib dose (21/7 dosing schedule) | 960

3. Primary Outcome: Maximum Plasma Concentration (Cmax) of Cobimetinib on Day 1, Cycle 1
Time Frame: Cycle 1: predose (0 hours [hr]) on Days 1, 2; 0.5, 1, 2, 4, 6 hr postdose on Day 1
Population: PK population included all participants who received study treatment and had at least one vemurafenib and cobimetinib plasma concentration available. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib: Participants received oral 60 mg cobimetinib QD on 21/7 dosing schedule and oral 720 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
- CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib: Participants received oral 60 mg cobimetinib QD on 21/7 dosing schedule and oral 960 mg vemurafenib BID on Days 1-28 of every cycle (1 Cycle=28 Days), until disease progression, unacceptable toxicity, or any other discontinuation criteria were met.
Arm/Group | DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 5 | 8 | 26 | 3 | 4 | 4 | 4 | 5 | 27 | 38
nanograms per milliliter (ng/mL) | 159 (110) | 146 (100) | 121 (96) | 136 (81) | 130 (53) | 133 (37) | 146 (79) | 93.6 (26) | 84.3 (67) | 105 (64)

4. Primary Outcome: Cmax of Cobimetinib on Day 1, Cycle 1 in Cohort 3
Time Frame: Cycle 1: predose (0 hr) on Days 1, 2; 0.5, 1, 2, 4, 6 hr postdose on Day 1
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 2
ng/mL | 51.6 (50.1)

5. Primary Outcome: Time Taken to Reach Maximum Plasma Concentration (Tmax) of Cobimetinib on Day 1, Cycle 1
Time Frame: Cycle 1: predose (0 hr) on Days 1, 2; 0.5, 1, 2, 4, 6 hr postdose on Day 1
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 5 | 8 | 26 | 3 | 4 | 4 | 4 | 2 | 5 | 27 | 38
hours | 4.00 [2.0 to 5.5] | 4.0 [2.0 to 27] | 4.00 [1.0 to 25] | 2.03 [2.0 to 24] | 3.99 [1.0 to 6.2] | 4.02 [4.0 to 4.1] | 4.03 [4.0 to 4.3] | 3.05 [2.0 to 4.1] | 4.00 [2.0 to 6.0] | 4.00 [0.5 to 6.0] | 4.00 [1.0 to 24]

6. Primary Outcome: Area Under Concentration Versus Time Curve (AUC) Over a Period of 24 Hours (AUC0-24) of Cobimetinib on Day 1, Cycle 1
Time Frame: Cycle 1: predose (0 hr) on Days 1, 2; 0.5, 1, 2, 4, 6 hr postdose on Day 1
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours per milliliter (ng*h/mL)
Arm/Group | DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 5 | 8 | 26 | 3 | 4 | 4 | 4 | 5 | 27 | 38
nanograms*hours per milliliter (ng*h/mL) | 2280 (90) | 1990 (99) | 1790 (88) | 1300 (35) | 1850 (35) | 1600 (29) | 2300 (100) | 1410 (29) | 1220 (63) | 1530 (65)

7. Primary Outcome: AUC0-24 of Cobimetinib on Day 1, Cycle 1 of Cohort 3
Time Frame: Cycle 1: predose (0 hr) on Days 1, 2; 0.5, 1, 2, 4, 6 hr postdose on Day 1
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 2
ng*h/mL | 727 (556)

8. Primary Outcome: Cmax of Cobimetinib on Day 14 (Steady State), Cycle 1
Time Frame: Cycle 1: predose (0 hr) on Days 8, 14; 0.5, 1, 2, 4, 6 hr postdose on Day 14
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 5 | 8 | 25 | 3 | 3 | 3 | 4 | 3 | 3 | 25 | 32
ng/mL | 342 (130) | 307 (75) | 232 (80) | 239 (14) | 414 (16) | 195 (48) | 383 (50) | 215 (19) | 350 (37) | 177 (74) | 200 (91)

9. Primary Outcome: Tmax of Cobimetinib on Day 14 (Steady State), Cycle 1
Time Frame: Cycle 1: predose (0 hr) on Days 8, 14; 0.5, 1, 2, 4, 6 hr postdose on Day 14
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 5 | 8 | 25 | 3 | 3 | 3 | 4 | 3 | 3 | 25 | 32
hours | 2.0 [0.98 to 4.0] | 3.98 [2.0 to 7.0] | 4.02 [0.5 to 8.0] | 4.00 [4.0 to 4.1] | 6.00 [4.9 to 6.1] | 6.0 [2.0 to 6.0] | 4.03 [2.2 to 6.1] | 4.08 [4.0 to 6.1] | 4.00 [3.9 to 4.1] | 4.04 [2.0 to 8.0] | 4.00 [0.0 to 8.0]

10. Primary Outcome: AUC0-24 of Cobimetinib on Day 14, Cycle 1
Time Frame: Cycle 1: predose (0 hr) on Days 8, 14; 0.5, 1, 2, 4, 6 hr postdose on Day 14
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 5 | 8 | 25 | 3 | 3 | 3 | 4 | 3 | 3 | 25 | 32
ng*h/mL | 5180 (170) | 4800 (76) | 3540 (83) | 4500 (17) | 7020 (27) | 3820 (48) | 6360 (46) | 3520 (35) | 5790 (36) | 2540 (84) | 3220 (124)

11. Primary Outcome: Clearance (CL) of Cobimetinib on Day 14 (Steady State), Cycle 1
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: Cycle 1: predose (0 hr) on Days 8, 14; 0.5, 1, 2, 4, 6 hr postdose on Day 14
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters per hour (L/h)
Arm/Group | DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 5 | 8 | 25 | 3 | 3 | 3 | 4 | 3 | 3 | 25 | 32
Liters per hour (L/h) | 11.6 (170) | 12.5 (76) | 17.0 (83) | 13.3 (17) | 8.55 (27) | 21.0 (48) | 15.7 (46) | 17.0 (35) | 13.8 (36) | 23.6 (84) | 18.6 (124)

12. Primary Outcome: Cmax of Vemurafenib on Day -1, Cycle 1 in Participants Previously Treated With Vemurafenib Prior to Enrollment Into This Study
Time Frame: Predose (0 hr) on Days -1, 1; 2, 4, 6, 8 hr postdose on Day -1
Population: PK population. Here, number of participants analyzed = participants who were previously treated with vemurafenib prior to enrollment into this study.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (mcg/mL)
Arm/Group | DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 5 | 6 | 8 | 3 | 3 | 1 | 15 | 19
micrograms per milliliter (mcg/mL) | 36.4 (58) | 34.3 (34) | 60.9 (32) | 56.0 (16) | 36.4 (19) | 48.2 (NA) — Geometric coefficient of variation is not applicable as only 1 participant had evaluable data. | 40.9 (110) | 48.6 (37)

13. Primary Outcome: Cmax of Vemurafenib on Day -1, Cycle 1 of Cohorts 1C and 2A in Participants Previously Treated With Vemurafenib Prior to Enrollment Into This Study
Time Frame: Predose (0 hr) on Day -1, 1; 2, 4, 6, 8 hr postdose on Day -1
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib
Number analyzed (Participants) | 2 | 2
mcg/mL | 38.8 (9.61) | 48.8 (35.4)

14. Primary Outcome: Tmax of Vemurafenib on Day -1, Cycle 1 in Participants Previously Treated With Vemurafenib Prior to Enrollment Into This Study
Time Frame: Predose (0 hr) on Day -1, 1; 2, 4, 6, 8 hr postdose on Day -1
Population: as for outcome 12
Measure: Median (Full Range); unit: hours
Arm/Group | DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 5 | 6 | 8 | 2 | 3 | 2 | 3 | 1 | 15 | 19
hours | 2.42 [1.3 to 4.5] | 2.50 [0.7 to 7.5] | 3.69 [1.1 to 11] | 4.55 [3.1 to 6.0] | 2.03 [0.9 to 2.5] | 1.65 [1.3 to 2.0] | 1.92 [0.6 to 4.8] | 0.83 [NA to NA] — Full range is not applicable as only 1 participant had evaluable data. | 2.33 [0.3 to 8.1] | 1.93 [0.6 to 7.5]

15. Primary Outcome: Cmax of Vemurafenib on Day 1, Cycle 1 in BRAFi-naïve Participants
Time Frame: Predose (0 hr) on Day 1, 2; 0.5, 1, 2, 4, 6 hr postdose on Day 1
Population: PK population.Here, number of participants analyzed = participants who were BRAFi-naïve participants.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 16 | 1 | 3 | 1 | 3 | 11 | 19
mcg/mL | 3.99 (73) | 2.31 (NA) — Geometric coefficient of variation is not applicable as only 1 participant had evaluable data. | 4.16 (78) | 1.25 (NA) — Geometric coefficient of variation is not applicable as only 1 participant had evaluable data. | 2.55 (170) | 2.60 (70) | 2.78 (57)

16. Primary Outcome: Cmax of Vemurafenib on Day 1, Cycle 1 in Cohort 1A in BRAFi-naïve Participants
Time Frame: Predose (0 hr) on Day 1, 2; 0.5, 1, 2, 4, 6 hr postdose on Day 1
Population: PK population. Here, number of participants analyzed = participants who were BRAFi-naïve participants.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib
Number analyzed (Participants) | 2
mcg/mL | 2.08 (1.64)

17. Primary Outcome: Tmax of Vemurafenib on Day 1, Cycle 1 in BRAFi-naïve Participants
Time Frame: Predose (0 hr) on Day 1, 2; 0.5, 1, 2, 4, 6 hr postdose on Day 1
Population: PK population. Here, number of participants analyzed = participants who were BRAFi-naïve participants.
Measure: Median (Full Range); unit: hours
Arm/Group | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 2 | 16 | 1 | 3 | 1 | 3 | 11 | 19
hours | 5.2 [4.4 to 6.0] | 4.15 [1.0 to 6.0] | 5.17 [NA to NA] — Full range is not applicable as only 1 participant had evaluable data. | 5.33 [2.0 to 6.2] | 2.08 [NA to NA] — Full range is not applicable as only 1 participant had evaluable data. | 4.00 [2.0 to 6.0] | 4.00 [2.0 to 6.0] | 4.00 [1.0 to 24]

18. Primary Outcome: Cmax of Vemurafenib on Day 14, Cycle 1
Time Frame: Predose (0 hr) on Days 14, 15; 0.5, 1, 2, 4, 6, 8 hr postdose on Day 14
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 5 | 8 | 25 | 3 | 3 | 3 | 4 | 3 | 3 | 25 | 32
mcg/mL | 34.7 (41) | 29.4 (25) | 43.7 (37) | 31.7 (42) | 51.3 (14) | 43.6 (45) | 30.6 (53) | 40.9 (20) | 33.7 (16) | 33.3 (58) | 36.3 (29)

19. Primary Outcome: Tmax of Vemurafenib on Day 14, Cycle 1
Time Frame: Predose (0 hr) on Days 14, 15; 0.5, 1, 2, 4, 6, 8 hr postdose on Day 14
Population: PK population. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Median (Full Range); unit: hours
Arm/Group | DES (Cohort 1): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 1C): 60 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 1D): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 2): 80 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 2A): 100 mg Cobimetinib + 720 mg Vemurafenib | DES (Cohort 3): 60 mg Cobimetinib + 960 mg Vemurafenib | DES (Cohort 4): 80 mg Cobimetinib + 960 mg Vemurafenib | CES (Cohort 1A): 60 mg Cobimetinib + 720 mg Vemurafenib | CES (Cohort 1B): 60 mg Cobimetinib + 960 mg Vemurafenib
Number analyzed (Participants) | 5 | 8 | 25 | 3 | 3 | 3 | 4 | 3 | 3 | 25 | 32
hours | 1.98 [0.0 to 7.7] | 2.15 [0.0 to 7.3] | 1.95 [0.0 to 8.0] | 1.98 [0.3 to 6.5] | 0.33 [0.2 to 8.2] | 5.6 [1.7 to 5.6] | 1.05 [0.0 to 6.4] | 1.83 [0.8 to 4.4] | 1.85 [0.1 to 4.0] | 1.17 [0.0 to 7.9] | 1.90 [0.0 to 7.6]

20. Secondary Outcome: Percentage of Participants With an Objective Response of Complete Response (CR) or Partial Response (PR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version (V) 1.1
Description: Tumor response of CR or PR is considered as objective response. CR: disappearance of all target lesions, reduction in short axis <10 millimeters in pathological lymph nodes (target and non-target lesions); PR: at least a 30 percent (%) decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter. Responses were confirmed by repeat assessments ≥4 weeks after initial documentation.
Time Frame: Assessed at screening (within 28 days prior to initiation of Cycle 1), every 6 weeks thereafter until disease progression (up to 82 months)
Population: Efficacy evaluable population who had measurable disease at baseline and had either a post-baseline tumour assessment or progressed before any tumour assessment was included in the analysis of this outcome.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vemurafenib PD Participants | BRAFi-naïve Participants
Number analyzed (Participants) | 66 | 63
percentage of participants | 15.2 [7.5 to 25.5] | 87.3 [76.7 to 94.4]

21. Secondary Outcome: Percentage of Participants With Disease Progression According to RECIST V 1.1
Description: Progressive disease (PD) according to RECIST V 1.1: at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study (nadir), including baseline; in addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm; appearance of 1 or more lesions is also considered as progression.
Time Frame: Assessed at screening (within 28 days prior to initiation of Cycle 1), every 6 weeks thereafter until disease progression or death (up to 82 months)
Population: as for outcome 20
Measure: Number; unit: percentage of participants
Arm/Group | Vemurafenib PD Participants | BRAFi-naïve Participants
Number analyzed (Participants) | 66 | 63
percentage of participants | 36.4 | 3.2

22. Secondary Outcome: Median Duration of Response (DOR)
Description: Duration of response, defined as the time from first occurrence of a documented objective response until the time of disease progression, as determined by investigator review of tumor assessments using RECIST v 1.1, or death from any cause during the study (that is within 30 days after the last dose of study treatment).
Time Frame: Time from first occurrence of objective response until the time of disease progression or death from any cause (up to 82 months)
Population: Efficacy evaluable population who had measurable disease at baseline and had either a post-baseline tumour assessment or progressed before any tumour assessment was included in the analysis of this outcome. Number of participants analysed who were evaluated for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vemurafenib PD Participants | BRAFi-naïve Participants
Number analyzed (Participants) | 10 | 55
months | 6.8 [4.9 to 10.4] | 14.3 [9.7 to 23]

23. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of randomization to the date of death due to any cause. Participants were censored at the last date of tumor measurement, the last date in the study drug log, or the date of last follow-up. OS analyzed using Kaplan-Meier estimate.
Time Frame: as for outcome 21
Population: as for outcome 20
Measure: Median (Full Range); unit: months
Arm/Group | Vemurafenib PD Participants | BRAFi-naïve Participants
Number analyzed (Participants) | 66 | 63
months | 8.5 [1.6 to 76.4] | 31.8 [2.7 to 69.2]

24. Secondary Outcome: Average Percent Change From Baseline in Fluorodeoxyglucose-positron Emission Tomography (FDG-PET) at Cycle 1 and Cycle 2
Description: The pharmacodynamic effect of cobimetinib in combination with vemurafenib was assessed by measuring changes in FDG uptake as characterized by the lean body mass corrected (LBM) maximum standardized uptake value (SUV max) measurement using FDG-PET. Post-baseline timepoint Cycle 1 was averaged between Days 10 to 14 and Cycle 2 for Days 14+7.
Time Frame: Cycle 1 (Days 10 to 14), Cycle 2 (Days 14+7)
Population: Safety evaluable population who received combination study treatment (Cobimetinib + Vemurafenib) was included in the analysis of this outcome. Here, number of participants analyzed = participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: Percent change in FDG-PET
Arm/Group | Vemurafenib PD Participants | BRAFi-naïve Participants
Number analyzed (Participants) | 63 | 63
Percent change in FDG-PET
  Baseline (n=63,63) | 8.75 (5.55) | 8.19 (5.00)
  Percent Change at Cycle 1 (Days 10-14) (n=59,60): number analyzed (Participants) | 59 | 60
  Percent Change at Cycle 1 (Days 10-14) (n=59,60) | -43.33 (26.00) | -65.74 (14.82)
  Percent Change at Cycle 2 (Days 14+7) (n=50,56): number analyzed (Participants) | 50 | 56
  Percent Change at Cycle 2 (Days 14+7) (n=50,56) | -33.09 (35.18) | -70.73 (17.05)

25. Secondary Outcome: Pharmacodynamics: Number of Participants With Mitogen-Activated Protein Kinase (MAPK) Inhibition, as Assessed by Immunohistochemistry (IHC)
Description: Changes in effector molecules of the MAPK pathway that are directly or indirectly affected by BRAF and MEK inhibition (including but not limited to ERK and phosphorylated ERK and MEK) by IHC using biopsies at baseline, between Days 10-14 of Cycle 1, and at disease progression. IHC is a staining process performed on fresh/frozen tumor tissue samples.
Time Frame: At baseline; Cycle 1: Day 14; at disease progression (Up to 32 months)
Population: Number of participants analyzed=number of participants available for analysis of this outcome measure.
Measure: Number; unit: participants
Arm/Group | Vemurafenib PD Participants | BRAFi-naïve Participants
Number analyzed (Participants) | 7 | 5
participants | 7 | 5

ADVERSE EVENTS:
Time Frame: Up to 82 months
Description: Safety data was not reported per dose/regimen cohort. Due to final analysis data for adverse events were reported collectively for both the reporting groups- Vemurafenib PD and BRAFi-naïve participants along with Cobimetinib Monotherapy. Data is presented based on the final CSR. As of 2017 per-cohort data were not collected.
Arm/Group | Vemurafenib PD Participants | BRAFi-naïve Participants | Cobimetinib Monotherapy (100 mg or 60 mg)
Serious Adverse Events (participants affected / at risk) | 21/66 | 36/63 | 0/2
Other Adverse Events (participants affected / at risk) | 64/66 | 63/63 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib PD Participants (N=66) | BRAFi-naïve Participants (N=63) | Cobimetinib Monotherapy (100 mg or 60 mg) (N=2)
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0
Iridocyclitis (Eye disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0
Biloma (Hepatobiliary disorders) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1 | 0
Pneumonia chlamydial (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 7 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Vogt-koyanagi-harada syndrome (Eye disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Face Oedema (General disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0
Haemtemesis (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Hypersenstivity (Immune system disorders) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 4 | 0
Streptococcal bacteraemia (Infections and infestations) | 0 | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Glomerulonephritis (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1 | 0
Chorioretinopathy (Eye disorders) | 0 | 1 | 0
Uveitis (Eye disorders) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Seizure (Nervous system disorders) | 1 | 5 | 0
Brain oedema (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Salpingo-Oophorectomy unilateral (Surgical and medical procedures) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib PD Participants (N=66) | BRAFi-naïve Participants (N=63) | Cobimetinib Monotherapy (100 mg or 60 mg) (N=2)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 12 | 44 | 0
Rash (Skin and subcutaneous tissue disorders) | 18 | 33 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 19 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 | 22 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 17 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 16 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 7 | 9 | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 | 10 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 3 | 19 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 20 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 9 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 7 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 | 7 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 5 | 0
Acne (Skin and subcutaneous tissue disorders) | 2 | 4 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 2 | 5 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 6 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 2 | 5 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 1 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 2 | 4 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 31 | 52 | 2
Nausea (Gastrointestinal disorders) | 22 | 37 | 1
Vomiting (Gastrointestinal disorders) | 13 | 30 | 1
Abdominal pain (Gastrointestinal disorders) | 10 | 13 | 1
Constipation (Gastrointestinal disorders) | 10 | 13 | 1
Abdominal distension (Gastrointestinal disorders) | 6 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 4 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 8 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 0
Ascites (Gastrointestinal disorders) | 4 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 5 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 4 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 9 | 0
Fatigue (General disorders) | 18 | 46 | 1
Oedema peripheral (General disorders) | 11 | 27 | 1
Pyrexia (General disorders) | 11 | 27 | 0
Chills (General disorders) | 10 | 17 | 1
Mucosal inflammation (General disorders) | 3 | 5 | 1
Asthenia (General disorders) | 5 | 2 | 0
Chest pain (General disorders) | 2 | 5 | 0
Malaise (General disorders) | 2 | 5 | 0
Influenza like illness (General disorders) | 1 | 6 | 0
Blood alkaline phophatase increased (Investigations) | 10 | 22 | 1
Blood creatine phosphokinase increased (Investigations) | 10 | 30 | 1
Aspartate aminotransferase increased (Investigations) | 6 | 22 | 0
Alanine aminotransferase increased (Investigations) | 4 | 25 | 0
Blood creatinine increased (Investigations) | 6 | 21 | 0
Blood bilirubin increased (Investigations) | 6 | 9 | 0
Electrocardiogram QT prolonged (Investigations) | 4 | 5 | 0
Weight decreased (Investigations) | 3 | 4 | 0
Gamma-glutamyl transferase increased (Investigations) | 1 | 8 | 0
Lymphocyte count decreased (Investigations) | 3 | 7 | 0
Blood uric acid increased (Investigations) | 0 | 4 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 31 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 20 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 11 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 7 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 4 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 5 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0
Decreased appetite (Metabolism and nutrition disorders) | 14 | 17 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 16 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 4 | 8 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 9 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 8 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 4 | 5 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 10 | 0
Headache (Nervous system disorders) | 13 | 19 | 0
Dizziness (Nervous system disorders) | 9 | 9 | 0
Paraesthesia (Nervous system disorders) | 5 | 4 | 0
Dysgeusia (Nervous system disorders) | 2 | 8 | 0
Memory impairment (Nervous system disorders) | 0 | 4 | 0
Sunburn (Injury, poisoning and procedural complications) | 13 | 23 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 13 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 16 | 0
Folliculitis (Infections and infestations) | 0 | 7 | 1
Urinary tract infection (Infections and infestations) | 3 | 6 | 0
Nasopharyngitis (Infections and infestations) | 1 | 4 | 0
Sinusitis (Infections and infestations) | 0 | 6 | 0
Vision blurred (Eye disorders) | 2 | 14 | 0
Photophobia (Eye disorders) | 2 | 5 | 0
Visual impairment (Eye disorders) | 4 | 6 | 0
Lacrimation increased (Eye disorders) | 1 | 4 | 0
Anaemia (Blood and lymphatic system disorders) | 11 | 23 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 6 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 0
Depression (Psychiatric disorders) | 4 | 5 | 0
Anxiety (Psychiatric disorders) | 3 | 7 | 0
Insomnia (Psychiatric disorders) | 3 | 8 | 0
Hypertension (Vascular disorders) | 6 | 18 | 1
Lymphoedema (Vascular disorders) | 0 | 6 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 15 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 15 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 11 | 1
Transaminases increased (Investigations) | 0 | 4 | 1
Weight increased (Investigations) | 0 | 4 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4 | 0
Peripheral swelling (General disorders) | 3 | 5 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 13 | 0
Seizure (Nervous system disorders) | 0 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT01271803/Prot_SAP_000.pdf